CLINICAL TRIAL: NCT02043652
Title: Efficacy of Chloroquine and Primaquine for the Treatment of Plasmodium Vivax Malaria in Cruzeiro do Sul, Acre, Brazil
Brief Title: Plasmodium Vivax Efficacy Trial in Cruzeiro do Sul, Acre, Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-CGH-6371
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2014-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chloroquine and primaquine (Experimental): Patients will receive 3-day treatment with chloroquine and 7-day treatment with primaquine in accordance to treatment guidelines in Brazil for P vivax malaria. All patients will receive the same treatment as there is no comparison arm.
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Chloroquine — Patients will receive 3-day treatment with chloroquine in accordance to treatment guidelines in Brazil. All patients will receive the same treatment as there is no comparison arm.
Drug: Primaquine — Patients will receive 7-day treatment with primaquine, in conjunction with chloroquine, in accordance to treatment guidelines in Brazil. All patients will receive the same treatment as there is no comparison arm.

SUMMARY:
Background: The World Health Organization recommends that antimalarial treatment policies be evaluated every few years to check their efficacy. P. vivax malaria is the most common species in Brazil and cases are concentrated in the Amazon Region in Brazil.

Objectives: Assess the efficacy of chloroquine and primaquine for the treatment of P. vivax infections in Cruzeiro do Sul, Acre, Brazil.

Methods: An in vivo drug efficacy study will be conducted in Cruzeiro do Sul, Acre State, Brazil. At least 117 study participants ≥5 years of age with parasitologically confirmed P. vivax monoinfections will be treated under supervision with chloroquine (CQ) for three days at a daily dose of approximately 25 mg/Kg in accordance with the Brazilian National Malaria Control guidelines. For patients with normal glucose 6 phosphate dehydrogenase activity levels, investigators will add primaquine at dose of 0.5mg/Kg per day for 7 days. Clinical and parasitologic parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy and for a total period of 168 days (6 months) to evaluate chances of recrudescence, relapse, or reinfection. Blood samples will be taken to measure the CQ levels in blood on Day 7 and day of failure, if occurring in the initial 28 days of follow up. In addition, a blood sample will be collected on filter paper on first day and on day of suspected failure to help differentiate parasite genotypes using techniques based on polymerase chain reaction. Results from this drug efficacy study will be used to assist the Brazilian Ministry of Health in assessing their national malaria treatment policy for P. vivax malaria.

DETAILED DESCRIPTION:
Background The impact of malaria on the health and economic development of human populations is greatest in the tropics and subtropics. The World Health Organization (WHO) has estimated 216 million episodes of malaria in 2010, of which 174 million (81%) were in Africa. There were a total of 655,000 malaria deaths worldwide, approximately 86% of which in children under 5 years of age (WHO 2011). Although the majority of deaths occur among children in sub-Saharan Africa, malaria accounts for considerable morbidity in the Americas, particularly in the Amazon Basin.

Most countries in the Americas have adopted the WHO Global Strategy for Malaria Control, which relies on prompt and effective antimalarial treatment as the major means of reducing malaria morbidity and mortality (WHO 2008). The ultimate success of this strategy rests on the ability of ministries of health to provide antimalarial drugs with proven efficacy. Although a wide variety of methods have been used to assess resistance to antimalarial drugs in vivo methods, in vitro drug sensitivity testing, and molecular analyses, most national malaria control programs rely on data from in vivo efficacy trials to assess the efficacy of the current first- and second-line drugs and to decide if charges in malaria treatment policy are needed.

The most widely used approach to conduct in vivo drug efficacy trials in the Americas follows the guidelines of the WHO (WHO 2009) with the modifications recommended by the Pan American Health Organization for studies in the Americas (PAHO 2003). The goal of such studies is to assess antimalarial drugs currently being used for first-line treatment of uncomplicated malaria. Much of the effort to monitor antimalarial efficacy in the Americas has been done as part of the Amazon Network of Antimalarial Resistance Monitoring and the Amazon Malaria Initiative (PAHO 2012). This information is critical for guiding the development of rational antimalarial drug policies in endemic areas.

Chloroquine-resistant P. vivax was first reported from Papua New Guinea in 1989 in two Australian soldiers (Rieckmann, Davis et al. 1989). In 1995, a study in Irian Jaya, Indonesia showed resistance in at least 44% of the P. vivax patients treated with chloroquine (CQ) (Baird, Basri et al. 1995). Several investigators have reported cases of CQ-resistant P. vivax in South America. In 1996, in Guyana, Phillips et al. reported three patients in whom 25 mg/kg of CQ failed to eliminate parasitemia despite adequate therapeutic blood levels of CQ (Phillips, Keystone et al. 1996). Three years later, in the Brazilian Amazon region, Alecrim et al. reported a 12-year old girl with P. vivax malaria who continued to have parasitemia after receiving a supervised course of 25mg/kg of CQ (Alecrim, Alecrim et al. 1999). More recently, Soto et al. reported three cases of CQ-resistant P. vivax in Colombia (Soto, Toledo et al. 2001). In these last two studies, CQ blood levels were not measured and it is not possible to confirm that adequate therapeutic levels were achieved.

Because of the serious public health implications of CQ-resistant P. vivax in the Americas, it is critically important to limit reports to well-confirmed cases. In most cases, this will require measurement of CQ blood levels and genotyping of parasites from the initial infection and any suspected recrudescence. P. falciparum in vivo trials take advantage of well-established molecular markers that help differentiate cases of recrudescence and reinfection, by polymerase chain reaction (PCR) techniques. Although no universally accepted technique for this purpose exists for P. vivax, investigators plan to use the microsatellites, base pair repeats in the parasite genome, described by Imwong et al (Imwong, Sudimack et al. 2006). Investigators believe that having PCR-corrected analysis is especially important in the context of the long follow-up period, six months, investigators aim for this study.

Many malaria cases in the Americas are reported in Brazil (Silveira 2001; Oliveira-Ferreira, Lacerda et al. 2010). In 2011, 293,701 malaria cases were reported to the Brazilian National Reportable Disease Information System. Most of these cases (99.7%) occurred in the Amazon region, which encompasses the states of Acre, Amazonas, Amapa, Para, Maranhao, Mato Grosso, Roraima, Rondonia, and Tocantins. In this region, socio-economic and environmental conditions, such as presence of natural breeding sites and abundance of Anopheles mosquitoes, favor malaria transmission. Amazonas, Rondonia, Para, and Acre states were responsible for 85.5% of malaria cases in 2011 according to the Brazilian National Reportable Disease Information System. As in other regions of the world, malaria is seasonal in Brazil, cases increase during or after the rainy season (Costa 2009).

In 2011, 87,6% of malaria cases in Brazil were due to P. vivax alone, 11,3% to P. falciparum alone, and approximately 1.1% due to mixed infections with these two species. P. malariae is rarely seen in Brazil. Acre state saw a huge increase in malaria cases from 2003 to 2004 and from 2004 to 2005, 153% and 63%, respectively(Cesario and Cesario 2006). The Acre municipalities of Cruzeiro do Sul, Rodrigues Alves, and Mancio Lima municipalities were responsible for 67.7% of malaria cases in the state in 2006, when a malaria epidemic took place in this region. Table 1 shows the absolute number of malaria cases in Brazil and Acre state and their respective annual parasitologic index (API), which is the number of positive malaria slides per 1,000 residents per year.

Although currently there is no evidence of CQ-resistant P. vivax in Cruzeiro do Sul, Acre State, Brazil, the Ministry of Health would like to assess the efficacy of CQ and primaquine for the treatment of uncomplicated P. vivax malaria as part their effort to study antimalarial drug resistance within the country. This practice is in accordance with current WHO recommendations (WHO 2009).

Objectives

* To assess the therapeutic efficacy of CQ and primaquine for the treatment of P. vivax malaria in Cruzeiro do Sul, Acre State, Brazil.
* Estimate recrudescence and reinfection rates of P. vivax infection after parasite clearance with CQ and primaquine.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥5 years; Body weight <120 kg ; documented fever (axillary temperature >37.5o C) or history of fever during the previous 48 hours in the absence of another obvious cause of fever, such as pneumonia, otitis media, etc ; Monoinfection with P. vivax with parasitemia between 250 and 100,000 asexual parasites/µl as determined by microscopic examination of thick and thin peripheral blood smears ; Informed consent from the patient or parent/guardian (for those <18 years), assent from child (ages 7 to 17 years inclusive), patients 5 through 6 years old will not need an assent ; Willingness on the part of the patient to return to the clinic and/or receive home visits for regular check-ups during the 6-month (168 days) follow-up period ; Place of residence within 30-45 minutes of study site.

Exclusion Criteria:

* 1. Presence of malaria danger signs ; presence of other underlying chronic or severe diseases (e.g., cardiac, renal, hepatic diseases, HIV/AIDS, tuberculosis, malnutrition) ; History of hypersensitivity reactions to any of the drugs being tested ; Current pregnancy (either self-reported being pregnant at enrollment or a positive urine pregnancy test at time of enrollment), previous pregnancy is not an exclusion criteria

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Macedo de Oliveira, MD, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Hospital do Jurua, Cruzeiro do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroquine and Primaquine
Started (We corrected the information in the patient flow section.) | 119
Completed | 93
Not Completed | 26

BASELINE CHARACTERISTICS:
Groups:
- Chlorquine and Primaquine: Patients will receive 3-day treatment with chloroquine and 7-day treatment with primaquine in accordance to treatment guidelines in Brazil for P vivax malaria. All patients will receive the same treatment as there is no comparison arm.
  Chloroquine: Patients will receive 3-day treatment with chloroquine in accordance to treatment guidelines in Brazil. All patients will receive the same treatment as there is no comparison arm.
  Primaquine: Patients will receive 7-day treatment with primaquine, in conjunction with chloroquine, in accordance to treatment guidelines in Brazil. All patients will receive the same treatment as there is no comparison arm.
Arm/Group | Chlorquine and Primaquine
Number analyzed (Participants) | 119
Age, Continuous [Median (Full Range); unit: years] | 23.4 [5 to 67.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 65
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 119

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adequate Clearance of Parasites and Symptoms
Description: Investigators, according to WHO guidelines, will evaluate patients at regular intervals to evaluate symptom and parasitemia clearance.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorquine and Primaquine
Number analyzed (Participants) | 110
Participants | 110

2. Secondary Outcome: Number of Patients Reporting Relapses
Description: Evaluate the relapse rate, that is reappearance of parasites, for up to 6 months after treatment.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorquine and Primaquine
Number analyzed (Participants) | 119
Participants | 28

ADVERSE EVENTS:
Arm/Group | Chlorquine and Primaquine
Serious Adverse Events (participants affected / at risk) | 0/119
Other Adverse Events (participants affected / at risk) | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No